CLINICAL TRIAL: NCT07320209
Title: Investigation of Physiological and Neurocognitive Responses to Multisensory Food Cues in an Virtual Reality Environment
Brief Title: Physiological and Neurocognitive Responses to Multisensory Food Cues in VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zehra Margot Celik, Dr., Marmara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09.2025.25-0627
Record Dates: First submitted 2025-12-03; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Food cue; human-computer interaction; food craving; salivary composition; EEG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer Participants (Experimental): Participants will be exposed to real, virtual, and multisensory food cues, and their food craving levels, saliva composition, blood glucose, EEG activity, and body temperature will be measured. Salivary alpha-amylase will be analysed as a biomarker of physiological arousal during food cue exposure. University students aged 18 and older will participate in the study.
  Interventions: Behavioral: Real food; Behavioral: Virtual Reality Food

INTERVENTIONS:
Behavioral: Real food — Participants will be exposed to real foods and their food craving levels, saliva composition, blood glucose, EEG activity, and body temperature will be measured. Salivary alpha-amylase will be analysed as a biomarker of physiological arousal during food cue exposure.
Behavioral: Virtual Reality Food — Participants will be exposed to vitrual foods and their food craving levels, saliva composition, blood glucose, EEG activity, and body temperature will be measured. Salivary alpha-amylase will be analyse

SUMMARY:
This study aims to investigate how food cravings change when visual food cues are enriched with sound, smell, and interactive experiences in a virtual reality (VR) environment. A total of 34 healthy Marmara University students aged 18 and older will participate in the study between November 2025 and March 2026, with a possible extension until September 2026.

Participants will be exposed to real, virtual, and multisensory food cues, and their food craving levels, saliva composition, blood glucose, EEG activity, and body temperature will be measured. Salivary alpha-amylase will be analysed as a biomarker of physiological arousal during food cue exposure.

The study aims to compare how virtual food cues affect food craving and physiological responses compared to real food cues. Findings are expected to contribute to understanding eating behaviour, developing VR-based interventions for healthy nutrition, and encouraging interdisciplinary collaboration between nutrition and engineering fields.

DETAILED DESCRIPTION:
This study aims to fill an important gap in the literature by examining the extent to which food craving responses can be enhanced by incorporating not only visual cues but also auditory, olfactory, and food-interaction-based experiences within a VR environment. Furthermore, by utilising objective biological indicators such as changes in saliva composition, blood glucose levels, and EEG recordings, the study aims to analyse VR-based food cue exposure not only through subjective assessments but also through objective data. In this respect, the study is expected to provide original contributions both conceptually and methodologically by enabling a deeper understanding of the mechanisms that increase food cravings and the modulation of these processes through VR technologies. The findings will provide a scientific basis for the development of therapeutic VR interventions to regulate food cravings in the future.

The original value of the study lies in the comprehensive monitoring of the effect of multi-sensory food cues presented in a VR environment on food cravings in individuals using physiological (saliva secretion and composition, blood glucose level) and neurocognitive (EEG recordings) measurements, and evaluating them comparatively with the responses to the same cues in a real environment. Although the effect of real-world food cues on food cravings has been studied in detail in the literature, the extent to which similar multi-sensory cues in VR environments trigger such responses has not yet been sufficiently clarified. Furthermore, studies investigating the effects of integrating additional sensory elements such as smell and food sounds to enhance presence in VR environments are quite limited.

This study will include a total of 34 healthy volunteers (both female and male) aged 18 and over, selected from among Marmara University students between November 2025 and March 2026, who meet the inclusion criteria for the study. Ethical approval for conducting the study was obtained from the Marmara University Faculty of Medicine Ethics Committee for Non-Drug and Non-Medical Device Research. The sample size was calculated using the G*Power 3.1 programme, based on the t-test for dependent samples. The calculations were based on a medium effect size (Cohen's d = 0.5), 80% statistical power, and a 5% significance level (α = 0.05). According to the power analysis performed based on these parameters, it was predicted that statistically significant results could be achieved with at least 34 participants in the study. Taking into account possible data losses, it was decided to invite 41 individuals, which is 20% more than the sample size. Considering the limited number of EEG devices and the time required for each experimental condition, the sample size was determined based on both scientific reasons and practical possibilities. The experimental procedure for each participant will be randomised using a Latin square design. If the targeted sample size cannot be achieved, the data collection process is planned to be extended until June 2026. Verbal and written informed consent will be obtained from all participants prior to the data collection process.

Whether participants meet the inclusion and exclusion criteria determined prior to the experimental procedure will be determined by the researcher using a pre-assessment form. Following the signing of the informed consent form, participants' anthropometric measurements will be taken; their body temperatures will be measured using a non-contact thermometer, and their blood glucose levels will be measured using an Accu-Chek glucometer. Subsequently, a demographic information form containing variables such as age and gender will be administered. Prior to the experiment, participants will be assessed on whether they have had any previous virtual reality (VR) experience and their level of liking for the foods that will be presented during the experiment (chocolate biscuits and pickles). This assessment will be conducted using a Visual Analogue Scale (VAS) scored on a scale of 0 (do not like at all) to 100 (like very much).

In this study, a within-subjects experimental design will be applied, and participants' food cravings in response to real, virtual, and multisensory (visual, auditory, olfactory, and interactive) food cues will be examined comparatively alongside their physiological (saliva, blood glucose) and neurocognitive (EEG) responses. Each experimental condition will last two minutes, during which EEG recordings will be taken and a total of four saliva samples will be collected from participants every 30 seconds. α-amylase levels will be determined from these samples. Following each condition, the instantaneous food craving level will be assessed using the Visual Analogue Scale (VAS); subsequently, the Excessive Food Craving Scale (EFCS) will be administered at the end of the food conditions.

Participants' body temperatures will be measured three times before, during, and after the experimental process to evaluate the effect of conditions experienced in the virtual reality environment on thermoregulation compared to real-world conditions. Thus, the potential effects of virtual environments on physiological responses, particularly in terms of body temperature, will be analysed comparatively. At the end of the experimental procedure, the Sense of Presence Scale (SPS) will be applied to assess participants' sense of presence in the virtual reality environment.

All data belonging to individuals participating in the study will be analysed using the SPSS 28.0 (Statistical Package for the Social Sciences for Windows) statistical package programme.

This research aims to yield social, academic, and economic benefits. The virtual reality (VR) applications developed within the scope of the project will contribute to improving individuals' quality of life by being used to understand and regulate nutritional behaviours in society. In particular, the development of interactive applications that increase awareness and consciousness regarding healthy eating will play an important role in reducing social problems related to nutrition. Academically, this study will encourage interdisciplinary collaborations (nutrition and dietetics - engineering) by offering methodological and theoretical innovations regarding the use of VR technologies in nutrition science, and will pave the way for the development of multidisciplinary master's theses. Thus, it will contribute to strengthening research capacity and training qualified researchers at national and international levels. Economically, the VR scenarios and measurement methods developed within the scope of the project have commercial application potential in the health technologies, food and nutrition sectors. The commercialisation of these applications will support the development of local software and technologies, enable the formation of new ventures (start-ups/spin-offs) in the health sector, and contribute to increasing competitiveness in the global market.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age.
* Individuals with a normal Body Mass Index according to the WHO classification.
* No known food allergies or eating disorder diagnoses.
* Voluntarily agree to participate in the study and sign an informed consent form.
* Be physically and psychologically suitable for virtual reality environment and electroencephalography (EEG) recording applications.

Exclusion Criteria:

* History of any neurological disease (e.g., epilepsy, vertigo) that may prevent the use of virtual reality goggles
* Allergy, intolerance, or sensitivity to foods used in the experimental procedure (e.g., chocolate biscuits, pickles)
* Significant loss or impairment of vision, hearing, or sense of smell.
* Sensitivity to the use of virtual reality devices (e.g. history of cyber sickness such as nausea, dizziness, etc.)
* Use of psychiatric medication, antidepressants, neuroleptics, or medication that may affect neurological status
* History of psychological conditions that may affect the working process, such as attention deficit, anxiety disorder, or panic attacks.
* Any discomfort in the salivary glands, insufficient saliva production, or dry mouth.
* Consumption of more than 21 units of alcohol per week (as this may affect food cravings and physiological parameters).
* History or diagnosis of abnormal brain electrical activity that may affect EEG measurements.
* History of substance dependence or any mental disorder that may affect cortical activity.
* Conditions that prevent body composition analysis (BIA) measurements (e.g. use of a pacemaker, limb amputation, lymphoedema, etc.).
* The presence of any language or cognitive barrier that prevents communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in EEG activation patterns in response to food cues | Baseline and peri-procedural (during exposure to food cues) within a single study session.
  Change in neural activation patterns measured by electroencephalography (EEG) in response to food cues presented in real-world and virtual reality environments. EEG data will be recorded using a 16-channel Brain Products LiveAmp system, assessing event-related potentials (P300, N200) and frequency band power (delta, theta, alpha, beta) across reward- and attention-related cortical regions.
Food craving questionnaire score | Baseline and immediately after completion of all experimental cue conditions within a single study session.
  Assesses subjective food craving responses using the Food Cravings Questionnaire-State (FCQ-S). Total scores range from 15 to 75, with higher scores indicating greater momentary food craving intensity.
Salivary α-amylase concentration (µU/mL) | Baseline and peri-procedural (during exposure to food cues) within a single study session.
  Salivary alpha-amylase concentration will be measured as an objective indicator of autonomic nervous system activation and physiological arousal in response to food cues presented in real-world and virtual reality environments.

SECONDARY OUTCOMES:
Salivary flow rate (mL/min) | Baseline and peri-procedural (during exposure to food cues) within a single study session.
  Salivary flow rate will be assessed as a physiological marker of appetitive and autonomic responses to food cues presented in real-world and virtual reality environments.
Capillary blood glucose level (mg/dL) | Measured pre-exposure and immediately post-exposure for each condition.
  Blood glucose changes will be used to assess metabolic reactivity to real and virtual food cues.
Subjective appetite rating score | Baseline and immediately after completion of each experimental cue condition within a single study session.
  Participants will rate their current desire to eat on a 0-100 mm Visual Analog Scale, where 0 = "no desire to eat" and 100 = "extreme desire to eat." Higher scores indicate greater craving intensity in response to food cues.
Body surface temperature (°C) | Baseline, during experimental cue exposure, and immediately post-exposure within a single study session.
  Body surface temperature will be measured as an indicator of autonomic physiological arousal and thermoregulatory responses during exposure to food cues presented in real-world and virtual reality environments.
Presence questionnaire score | Immediately after completion of all virtual reality experimental conditions within a single study session.
  Assesses the subjective sense of presence (the feeling of "being there") in the virtual environment using the Igroup Presence Questionnaire (IPQ). Total scores range from 0 to 6, with higher scores indicating a stronger sense of presence in the virtual environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) collected in this study will not be shared publicly. The data include sensitive physiological and neurocognitive measurements (EEG and salivary biomarkers) collected as part of a graduate thesis project. Data will be used solely for the purposes of the primary analyses described in the protocol and related scientific publications.